CLINICAL TRIAL: NCT02093702
Title: Impact of Structured Physical Activity Education Delivery on Hemoglobin A1c Levels, Blood Pressure, Lipid Profile, Body Mass Index, Waist Circumference, and Adherence to Canadian Diabetes Association Clinical Practice Guidelines Weekly Physical Activity Recommendations for Patients With Type 2 Diabetes Mellitus: A Pilot Study.
Brief Title: Impact of Structured Physical Activity Education Delivery in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Victoria Hospital, Canada (Other)
Responsible Party: Principal Investigator, Dr. Andrew Wozniak, MD, CCFP, Royal Victoria Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AW-100-SD
Record Dates: First submitted 2014-03-03; First posted 2014-03-21 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unstructured Physical Activity and Exercise Education Delivery (Active Comparator): 50 subjects will receive the standard approach to physical activity and exercise education from a Certified Diabetes Educator.
  Interventions: Behavioral: Unstructured Physical Activity and Exercise Education
- Structured Physical Activity and Exercise Education Delivery (Experimental): 50 subjects will receive physical activity and exercise education and behaviour counseling from a qualified Exercise Specialist (Registered Kinesiologist). These subjects will receive access to a community health and fitness centre as well as exercise instruction and on-going support and motivation from a YMCA Wellness Coach who focuses on establishing healthy behaviors towards the attainment of personal goals. Subjects will be requested to complete a lifestyle questionnaire at each appointment with their Wellness Coach. Subjects will receive a Physical Activity and Exercise Journal that will help them keep track of their weekly physical activity and exercise activities.
  Interventions: Behavioral: Physical activity and exercise education and behaviour counseling from a Registered Kinesiologist and a YMCA Wellness Coach

INTERVENTIONS:
Behavioral: Physical activity and exercise education and behaviour counseling from a Registered Kinesiologist and a YMCA Wellness Coach
  Arms: Structured Physical Activity and Exercise Education Delivery
Behavioral: Unstructured Physical Activity and Exercise Education
  Arms: Unstructured Physical Activity and Exercise Education Delivery

SUMMARY:
The objective of this study is to assess whether a structured exercise program compared to routine recommendation for exercise has any positive impact on disease outcome in patients with type 2 diabetes.

This study aims to assess whether a structured exercise program has an impact on the following determinants of the disease in type 2 diabetes: HbA1C, blood pressure, lipids, body mass index and waist circumference. It also aims to assess the compliance and retention of patients with type 2 diabetes in a structured exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman with type 2 diabetes
* Ready to begin regular physical activity
* Age equal to or greater than 18
* Age equal to or less than 64.

Exclusion Criteria:

* Any vascular disease
* Exhibits symptoms of coronary artery disease (CAD)
* History of losing balance because of dizziness
* History of losing consciousness
* Has a bone or joint problem that could be made worse by a change in physical activity
* Pregnant
* Has been excluded by the Patient's Physician for any other health-related reason not stated under these exclusion criteria.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Andrew Wozniak, MD, CCFP, Principal Investigator — Barrie and Community Family Health Team
Locations (1):
- Barrie and Community Family Health Team Diabetes Program, Barrie, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] J.R. Fowles, C. Shields, R.J.L. Murphy and P Dunbar. Developing Competency in Diabetes Education Volume 3: Physical Activity and Exercise Professional Resource Manual. The Canadian Diabetes Association. 2012. Toronto, Ontario. 110 pages.
- [Background] Canadian Diabetes Association Clinical Practice Guidelines Expert Committee; Booth G, Cheng AY. Canadian Diabetes Association 2013 clinical practice guidelines for the prevention and management of diabetes in Canada. Methods. Can J Diabetes. 2013 Apr;37 Suppl 1:S4-7. doi: 10.1016/j.jcjd.2013.01.010. Epub 2013 Mar 26. No abstract available. PMID 24070961
- [Background] Buse JB, Ginsberg HN, Bakris GL, Clark NG, Costa F, Eckel R, Fonseca V, Gerstein HC, Grundy S, Nesto RW, Pignone MP, Plutzky J, Porte D, Redberg R, Stitzel KF, Stone NJ; American Heart Association; American Diabetes Association. Primary prevention of cardiovascular diseases in people with diabetes mellitus: a scientific statement from the American Heart Association and the American Diabetes Association. Circulation. 2007 Jan 2;115(1):114-26. doi: 10.1161/CIRCULATIONAHA.106.179294. Epub 2006 Dec 27. PMID 17192512
- [Background] Gornall A, Levesque L, Sigal RJ. A Pilot Study of Physical Activity Education Delivery in Diabetes Education Centres in Ontario. Can J Diabetes. 2008;32(2):123-30. doi: 10.1016/S1499-2671(08)22009-5. Epub 2012 Dec 10. PMID 27056541
- [Background] Canadian Institute for Health Information. Pan-Canadian Primary Health Care Indicator Update Report. Canadian Institute for Health Information, 2012. Ottawa, Ontario. 198 pages.
- [Background] Chudyk A, Petrella RJ. Effects of exercise on cardiovascular risk factors in type 2 diabetes: a meta-analysis. Diabetes Care. 2011 May;34(5):1228-37. doi: 10.2337/dc10-1881. PMID 21525503
- [Background] Umpierre D, Ribeiro PA, Kramer CK, Leitao CB, Zucatti AT, Azevedo MJ, Gross JL, Ribeiro JP, Schaan BD. Physical activity advice only or structured exercise training and association with HbA1c levels in type 2 diabetes: a systematic review and meta-analysis. JAMA. 2011 May 4;305(17):1790-9. doi: 10.1001/jama.2011.576. PMID 21540423
- [Background] Plotnikoff RC, Taylor LM, Wilson PM, Courneya KS, Sigal RJ, Birkett N, Raine K, Svenson LW. Factors associated with physical activity in Canadian adults with diabetes. Med Sci Sports Exerc. 2006 Aug;38(8):1526-34. doi: 10.1249/01.mss.0000228937.86539.95. PMID 16888470
- [Background] McManus RM, Stitt LW, Bargh GJM. Population survey of diabetes knowledge and protective behaviours. Can J Diabetes. 2006;30:256-263.
- [Background] Majumdar SR, Johnson JA, Bowker SL, Booth GL, et al. A Canadian consensus for the standardized evaluation of quality improvement interventions in type 2 diabetes. Can J Diabetes. 2005 2005;29:220-229.
- [Background] McSweeney JC, Cody M, O'Sullivan P, Elberson K, Moser DK, Garvin BJ. Women's early warning symptoms of acute myocardial infarction. Circulation. 2003 Nov 25;108(21):2619-23. doi: 10.1161/01.CIR.0000097116.29625.7C. Epub 2003 Nov 3. PMID 14597589
- [Background] Zanuso S, Jimenez A, Pugliese G, Corigliano G, Balducci S. Exercise for the management of type 2 diabetes: a review of the evidence. Acta Diabetol. 2010 Mar;47(1):15-22. doi: 10.1007/s00592-009-0126-3. Epub 2009 Jun 3. PMID 19495557
- [Background] Kraus WE, Houmard JA, Duscha BD, Knetzger KJ, Wharton MB, McCartney JS, Bales CW, Henes S, Samsa GP, Otvos JD, Kulkarni KR, Slentz CA. Effects of the amount and intensity of exercise on plasma lipoproteins. N Engl J Med. 2002 Nov 7;347(19):1483-92. doi: 10.1056/NEJMoa020194. PMID 12421890
- [Background] Duncan GE, Perri MG, Theriaque DW, Hutson AD, Eckel RH, Stacpoole PW. Exercise training, without weight loss, increases insulin sensitivity and postheparin plasma lipase activity in previously sedentary adults. Diabetes Care. 2003 Mar;26(3):557-62. doi: 10.2337/diacare.26.3.557. PMID 12610001
- See also: YMCA Wellness Coaching — http://ymcaofsimcoemuskoka.ca/barrie-ymca-wellness-coaching/

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard PA Education for People With T2DM (From a CDE): Subjects in the control arm (n = 2) received the standard approach to PA education from a Canadian Certified Diabetes Educator (CDE).
- Structured PA Education Program for People With T2DM: Subjects in the experimental arm (n = 3) participated in a structured PA education program for people with T2DM.
Period: Overall Study
Arm/Group | Standard PA Education for People With T2DM (From a CDE) | Structured PA Education Program for People With T2DM
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard PA Education for People With T2DM (From a CDE) | Structured PA Education Program for People With T2DM | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin A1c (HbA1c) Levels
Time Frame: Baseline and 12 months
Measure: Mean (Full Range); unit: mmol/mol
Groups:
- Standard PA Education for People With T2DM (From a CDE): Group of subjects with Type 2 Diabetes Mellitus (T2DM) receiving physical activity (PA) education from a Certified Diabetes Educator (CDE).
- Structured PA Education Program for People With T2DM: Group of subjects with Type 2 Diabetes Mellitus (T2DM) receiving physical activity (PA) education from the Registered Kinesiologist and YMCA Wellness Coach.
Arm/Group | Standard PA Education for People With T2DM (From a CDE) | Structured PA Education Program for People With T2DM
Number analyzed (Participants) | 2 | 3
mmol/mol | 0.001 [0.0007 to 0.0013] | -0.007 [-0.0073 to -0.0067]

2. Primary Outcome: Mean Change in Systolic Blood Pressure
Time Frame: Baseline and 12 months
Measure: Mean (Full Range); unit: mm Hg
Arm/Group | Standard PA Education for People With T2DM (From a CDE) | Structured PA Education Program for People With T2DM
Number analyzed (Participants) | 2 | 3
mm Hg | 5.0 [2.0 to 7.0] | 7 [3 to 10]

3. Primary Outcome: Mean Change in Waist Circumference
Time Frame: Baseline and 12 months
Measure: Mean (Full Range); unit: cm
Groups:
- Structured PA Education Program for People With T2DM: Group of subjects with Type 2 Diabetes Mellitus (T2DM) receiving physical activity (PA) education from the Registered Kinesiologist and YMCA Wellness Coach.
  .
Arm/Group | Standard PA Education for People With T2DM (From a CDE) | Structured PA Education Program for People With T2DM
Number analyzed (Participants) | 2 | 3
cm | 0.7 [-1.5 to 3.7] | -3.4 [-4.8 to -2.0]

4. Primary Outcome: Mean Change in Body Mass Index
Time Frame: Baseline and 12 months
Measure: Mean (Full Range); unit: kg/m^2
Arm/Group | Standard PA Education for People With T2DM (From a CDE) | Structured PA Education Program for People With T2DM
Number analyzed (Participants) | 2 | 3
kg/m^2 | 0.6 [-1.2 to 1.8] | -2.0 [-2.8 to -1.0]

5. Primary Outcome: Mean Change in Serum Total Cholesterol
Time Frame: Baseline and 12 months
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | Standard PA Education for People With T2DM (From a CDE) | Structured PA Education Program for People With T2DM
Number analyzed (Participants) | 2 | 3
mmol/L | -0.75 [-0.87 to -0.62] | -0.13 [-0.17 to -0.10]

6. Primary Outcome: Mean Change in HDL-C
Time Frame: Baseline and 12 months
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | Standard PA Education for People With T2DM (From a CDE) | Structured PA Education Program for People With T2DM
Number analyzed (Participants) | 2 | 3
mmol/L | -0.03 [-0.05 to -0.01] | 0.08 [0.06 to 0.09]

7. Primary Outcome: Mean Change in LDL-C
Time Frame: Baseline and 12 months
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | Standard PA Education for People With T2DM (From a CDE) | Structured PA Education Program for People With T2DM
Number analyzed (Participants) | 2 | 3
mmol/L | -0.59 [-0.63 to -0.55] | 0.08 [0.063 to 0.095]

8. Primary Outcome: Mean Change in Triglycerides (TGs)
Time Frame: Baseline and 12 months
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | Standard PA Education for People With T2DM (From a CDE) | Structured PA Education Program for People With T2DM
Number analyzed (Participants) | 2 | 3
mmol/L | -0.28 [-0.46 to -0.10] | -0.63 [-0.71 to -0.57]

9. Primary Outcome: Mean Change in Total Cholesterol: HDL-C Ratio
Time Frame: Baseline and 12 months
Measure: Mean (Full Range); unit: mmol/L:mmol/L
Arm/Group | Standard PA Education for People With T2DM (From a CDE) | Structured PA Education Program for People With T2DM
Number analyzed (Participants) | 2 | 3
mmol/L:mmol/L | -0.7 [-0.87 to -0.53] | -0.4 [-0.5 to -0.3]

10. Primary Outcome: Mean Change in Diastolic Blood Pressure
Time Frame: Baseline and 12 months
Measure: Mean (Full Range); unit: mm Hg
Arm/Group | Standard PA Education for People With T2DM (From a CDE) | Structured PA Education Program for People With T2DM
Number analyzed (Participants) | 2 | 3
mm Hg | 5 [4 to 6] | 2 [-1 to 4]

11. Secondary Outcome: Mean Change in Adherence to the Canadian Diabetes Association's Clinical Practice Guidelines Aerobic Exercise Recommendations
Description: The Canadian Diabetes Association's Clinical Practice Guidelines recommends at least 150 minutes per week of aerobic exercise.
Time Frame: Baseline and 12 months
Measure: Mean (Full Range); unit: minutes/week
Arm/Group | Standard PA Education for People With T2DM (From a CDE) | Structured PA Education Program for People With T2DM
Number analyzed (Participants) | 2 | 3
minutes/week | 58 [20 to 96] | 26 [10 to 55]

12. Secondary Outcome: Mean Change in Adherence to the Canadian Diabetes Association's Clinical Practice Guidelines Resistance Exercise Recommendations
Description: The Canadian Diabetes Association's Clinical Practice Guidelines recommends at least 2 sessions per week of resistance exercise.
Time Frame: Baseline and 12 months
Measure: Mean (Full Range); unit: sessions/week
Arm/Group | Standard PA Education for People With T2DM (From a CDE) | Structured PA Education Program for People With T2DM
Number analyzed (Participants) | 2 | 3
sessions/week | 0 [-0.6 to 0.6] | 0.7 [0.5 to 1.1]

ADVERSE EVENTS:
Description: Serious and other [not including serious] adverse events were not monitored/assessed.
Groups:
- Standard PA Education for People With T2DM (From a CDE): Group of subjects receiving physical activity (PA) education from a Certified Diabetes Educator (CDE).
Arm/Group | Structured PA Education Program for People With T2DM | Standard PA Education for People With T2DM (From a CDE)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No